CLINICAL TRIAL: NCT01283906
Title: A Randomized, Double-blind Study to Evaluate the Efficacy of MuGard Mucoadhesive Oral Wound Rinse for the Amelioration of Oral Mucositis in Subjects Receiving Chemoradiation Therapy for the Treatment of Cancers of the Head and Neck
Brief Title: A Study to Evaluate the Efficacy of MuGard for the Amelioration of Oral Mucositis in Head and Neck Cancer Patients
Acronym: MuGard
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Access Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APC-10U1101
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Oral Mucositis
Keywords: Mucositis; Head and Neck Cancer; Squamous Cell Cancer; Chemotherapy; Radiation Therapy; Oral Rinse
MeSH Terms: conditions — Stomatitis; Mucositis; Head and Neck Neoplasms; Neoplasms, Squamous Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MuGard (Experimental): Mucoadhesive Oral Wound Rinse
  Interventions: Device: MuGard
- Control Rinse (Sham Comparator): Aqueous Control Rinse.
  Interventions: Device: Control Rinse

INTERVENTIONS:
Device: MuGard — Mucoadhesive Oral Wound Rinse. 5 mL oral rinse is used to cover the entire oral cavity every 3 hours (while awake) for up to a maximum of 6 doses per day
  Arms: MuGard
Device: Control Rinse — Aqueous Control Rinse. 5 mL oral rinse is used to cover the entire oral cavity every 3 hours (while awake) for up to a maximum of 6 doses per day.
  Arms: Control Rinse

SUMMARY:
This study is a randomized, double-blind, sham-controlled, two-arm study conducted in subjects receiving chemoradiation therapy for the treatment of head and neck cancer to assess the efficacy of MuGard. The study will evaluate the ability of MuGard to reduce the symptoms of oral mucositis. The study includes a treatment period of approximately 7 weeks depending on the subject's prescribed radiation plan.

MuGard is a liquid that is classified as a medical device. It is a hydrated polymer system (oral hydrogel) and is intended for the management of oral mucositis/stomatitis. When gently distributed within the mouth, the mucoadhesive formulation results in the formation of a protective coating over the oral mucosa. Subjects undergoing chemotherapy with radiation for the treatment of head and neck cancer are at high risk of developing oral mucositis as an adverse side-effect of cancer treatment. MuGard was previously shown to reduce the incidence and severity of mucositis in head and neck cancer patients undergoing radiation therapy when compared with data from historical control groups. The purpose of this study is to perform a direct comparison of the effectiveness of MuGard with a control group.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the study if they:

1. Are willing and able to understand and sign an informed consent form (ICF) for the study approved by the Investigator's local or a central Institutional Review Board (IRB) or Independent Ethics Committee (IEC)
2. Are males or females aged 18 years or older
3. Have recently-diagnosed, pathologically-confirmed cancer of the head and neck (e.g., oral cavity, oropharynx, hypopharynx, larynx; nasopharynx, lips, sinuses, salivary glands, or unknown primary)that will be treated with CRT (with or without induction therapy prior to CRT)
4. Have a plan to receive a continuous course of conventional external beam irradiation delivered as single daily fractions of 2.0 Gy to 2.2 Gy with a cumulative radiation dose between 50 Gy and 72 Gy with concomitant chemotherapy. Planned radiation treatment fields must include at least two oral sites (buccal mucosa, floor of mouth, tongue, soft palate) with each site receiving at least 50 Gy
5. Have Karnofsky performance score (KPS) >= 80% or Eastern Cooperative Oncology Group (ECOG) score of <= 1 (See Appendix B and C for KPS and ECOG scores respectively)
6. Have the ability to comply with the MuGard product insert

Exclusion Criteria:

Subjects will be excluded from participation in the study if they:

1. Have major surgical procedure or significant traumatic injury within 2 weeks prior to the initiation of RT or anticipation of need for major surgical procedure during the course of the study
2. Have active infectious disease excluding oral candidiasis
3. Have presence of oral mucositis
4. Have chronic immunosuppression
5. Have use of any investigational agent within 30 days of randomization
6. Are female subjects who are pregnant or breastfeeding
7. Have known allergies or intolerance to MuGard Mucoadhesive Oral Wound Rinse, its ingredients, or the ingredients used in the sham control. The ingredients which appear in either formulation are as follows: benzalkonium chloride, benzyl alcohol, carbopol 971P, citric acid, glycerin, polysorbate 60, phosphoric acid, purified Water, sodium bicarbonate, sodium chloride, sodium saccharin
8. Have inability to give informed consent or comply with study requirements
9. Are unwilling to or unable to complete the subject diary
10. Have any other condition or prior therapy that in the opinion of the Investigator would make the subject unsuitable for the study or unable to comply with follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of MuGard on reducing the symptoms of oral mucositis using an Oral Mucositis Daily Questionnaire (OMDQ) | 7 weeks
  To evaluate the efficacy of MuGard administered every 3 hours up to six times a day (while awake) over approximately 7 weeks in subjects with head and neck cancers receiving up to a maximum cumulative radiation dose of 72 Gray (Gy) compared to sham control on reducing the symptoms of oral mucositis [area-under-the-curve (AUC) of Oral Mucositis Daily Questionnaire (OMDQ) Mouth and Throat Soreness (MTS) Question 2].

SECONDARY OUTCOMES:
To evaluate the efficacy of MuGard on delaying the onset of oral mucositis symptoms and reducing the impact on health and resource outcomes. | Approximately 7 weeks
  To evaluate the efficacy of MuGard administered every 3 hours up to six times a day (while awake) in subjects with head and neck cancers receiving up to a maximum cumulative radiation dose of 72 Gy compared to sham control on delaying the onset of oral mucositis symptoms (OMDQ MTS Question 2) and reducing the impact on health and resource outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: William Wisbeck, MD, Principal Investigator — Providence Hospital - Pacific Campus; Flynn Cancer Center; Dimitrios Papadopoulos, MD, Principal Investigator — Vassar Brothers Medical Center
Locations (18):
- United States (18):
  - Ironwood Cancer and Research Centers, Mesa, Arizona
  - 21st Century Oncology TRC Headquarters, Scottsdale, Arizona
  - St. Joseph's Mercy Cancer Center- Hot Springs Radiation Oncology, Hot Springs, Arkansas
  - Enloe Medical Center- Cancer Center, Chico, California
  - John Muir Medical Center, Concord, California
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Signature Healthcare Brockton Hospital, Brockton, Massachusetts
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - VA Western New York Health System, Buffalo, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - CaroMont Health Comprehensive Cancer Center, Gastonia, North Carolina
  - 21st Century Oncology- Carolina Radiation Medicine, Greenville, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - PeaceHealth St. Joseph Cancer Center, Bellingham, Washington
  - Providence Hospital - Pacific Campus; Flynn Cancer Center, Everett, Washington
  - Columbia St. Mary's Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Allison RR, Ambrad AA, Arshoun Y, Carmel RJ, Ciuba DF, Feldman E, Finkelstein SE, Gandhavadi R, Heron DE, Lane SC, Longo JM, Meakin C, Papadopoulos D, Pruitt DE, Steinbrenner LM, Taylor MA, Wisbeck WM, Yuh GE, Nowotnik DP, Sonis ST. Multi-institutional, randomized, double-blind, placebo-controlled trial to assess the efficacy of a mucoadhesive hydrogel (MuGard) in mitigating oral mucositis symptoms in patients being treated with chemoradiation therapy for cancers of the head and neck. Cancer. 2014 May 1;120(9):1433-40. doi: 10.1002/cncr.28553. PMID 24877167